CLINICAL TRIAL: NCT06610981
Title: Impact of Laser Acupuncture on Pain, Range of Motion and Function in Patients With Patellofemoral Pain Syndrome: A Randomized Sham-Controlled Trial
Brief Title: Laser Acupuncture on Pain, Range of Motion and Function in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Approval No. 2024-82
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: laser acuouncture; function; pain; range of motion
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Laser acupuncture group) (Experimental): Participants will receive Laser acupuncture with energy of 4 J per point for 80 s, with a total dosage of 24 J in each session, 2 times /week for 4 weeks. Additionally, traditional physical therapy program will be conducted to participants in the study group.
  Interventions: Device: Laser acupuncture; Other: traditional physical therapy
- Group B (Sham-laser acupuncture group) (Sham Comparator): Participants will receive the same intervention while the device turned off, in addition to the exercise program consisted of stretching for hamstring, gastrocnemius and iliotibial band, and strengthening exercises, which include isometric quadriceps exercises, straight leg raising, lateral straight leg raise, isometric hip adduction and squat to 30° knee flexion, 2 times /week for 4 weeks.
  Interventions: Other: traditional physical therapy; Device: Sham laser acupuncture

INTERVENTIONS:
Device: Laser acupuncture — Laser acupuncture will be used in this study with energy of 4 J per point for 80 s, with a total dosage of 24 J in each session, 2 times /week for 4 weeks
  Arms: Group A (Laser acupuncture group)
Other: traditional physical therapy — exercise program consisted of stretching for hamstring, gastrocnemius and iliotibial band, and strengthening exercises, which include isometric quadriceps exercises, straight leg raising, lateral straight leg raise, isometric hip adduction and squat to 30° knee flexion, 2 times /week for 4 weeks
Device: Sham laser acupuncture — Participants will receive laser acupuncture while the device is turned off.
  Arms: Group B (Sham-laser acupuncture group)

SUMMARY:
Patellofemoral pain syndrome (PFPS) is among the most prevalent forms of knee discomfort. The main complaint is typically anterior knee pain, which gets worse while jumping, bending knee, going up or down stairs, or sitting for long periods of time with bent knee. Teens and early adulthood are commonly affected by patellofemoral pain syndrome, with a higher frequency in females. In healthy general populations, the prevalence of patellofemoral pain syndrome is 22.7%, and in teens, it is 28.9%.

DETAILED DESCRIPTION:
The treatment goals of patellofemoral pain syndrome are to reduce pain, increase muscle strength, increase flexibility, and correct the patellar movement tract. Conservative methods should be used before invasive methods when treating PFPS. One of the ways that people with PFPS may benefit from improved knee function and long-term pain reduction is by strengthening their quadriceps muscles, which primarily reduce force in the patellofemoral joint. Conservative methods described in the literature include the following: modifying activities; electrophysical modalities like biofeedback; therapeutic ultrasound; neuromuscular electrical stimulation; thermotherapy; interferential current; transcutaneous electrical nerve stimulation (TENS); knee braces; strengthening the hamstring, anterior tibialis, and gluteal muscles; stretching for iliotibial band and lateral retinaculum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with patellofemoral pain syndrome (positive Clarkes sign and Waldron test)
* Age from 18 to 25 years
* Patients suffering from pain which aggravated by prolonged sitting, stair climbing, running, squatting, kneeling, hopping\jumping, overuse activities and relieved by rest for at least 3 months
* Visual analog scale (VAS) greater than 3 points in daily activity
* The ability to participate in the study and follow the treatment schedule.

Exclusion Criteria:

* Physiotherapy in the last 12 months
* Intra-articular injection in the last 3 months
* Other knee disorders such as: (osteoarthritis, previous knee surgery, history of knee arthroplasty, or traumatic injury related joint deformity)
* BMI greater than or equal 30
* Pregnancy
* Pacemaker insertion
* Photosensitivity
* History of using oral analgesic or NSAIDs in the previous 4 weeks,
* History of malignancy, psychiatric disorder, mental retardation, neurologic dysfunction, diabetes mellitus, or uncontrolled hypertension.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 4 weeks
  The visual analogue scale represents the pain range that a patient thinks they might experience. The line is typically 10 centimetres long, with or without markings at each centimetre serves as a representation of the range. The worst pain the patient could possibly envision is represented by one end, while; no pain; is represented by the other. The patient marks the scale by drawing a line on it to indicate the amount of discomfort they are experiencing from 0-10. Higher scores represent worse pain.

SECONDARY OUTCOMES:
Range of motion for knee flexion | 4 weeks
  A universal goniometer was used to assess knee flexion while the subject was lying prone. It is an accurate and trustworthy measuring device. It was assessed while resting prone and with the knee extended. While keeping the other foot in touch with the plinth, the patient was instructed to bring the heel of the leg being tested as near to the buttock as feasible. With one arm aligned with the lateral malleolus and the other with the greater trochanter, the fulcrum of the goniometry is situated on the lateral epicondyle of the examined knee. A range of motion of knee flexion ranged from 0-135°. The higher the range, the better the results.
Function of knee joint | 4 weeks
  A scale known as Kujala patellofemoral score will be used for assessment of the function of the patellofemoral pain syndrome. The scores of this rating system vary from 100 (a normal, painless, totally functional knee) to 0 (severe pain and dysfunction in the knee). Haddad et al. conducted research on the validity and reliability of the Arabic version of the scale. The greater the scores, the better the results.
Range of motion for knee extension | 4 weeks
  The dominant limbs hip and knee were bent to a 90-degree angle for the first assessment, while the foot was kept in a relaxed position. Knee extension, as demonstrated by Norkin &White with the universal goniometer. The normal ROM for knee extension is 135- 0º. Each person's knee extension range of motion was assessed three times, and the computations employed the arithmetic mean of the three measures. The lower the range, the better the results.

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Ali Hamada, PhD, Study Director — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Giza Governorate, Egypt

REFERENCES:
- [Derived] Allam NM, Alsirhani H, Alruwaili MB, Dosh DM, Alruwaili HM, Almazyad WH, Toson RA, Elimy DA, El-Sherbiny M, Ibrahim AM, Ebrahim HA, Nosseir N, Eladl MA, Ali ZA. Effect of laser acupuncture on pain, range of motion, and function in patellofemoral pain syndrome: a randomised controlled trial. Front Med (Lausanne). 2025 Jul 15;12:1613197. doi: 10.3389/fmed.2025.1613197. eCollection 2025. PMID 40735438